CLINICAL TRIAL: NCT05703152
Title: Effect of a Combined Therapeutic Exercise Program on Neuropathic Pain and Perceived Quality of Life in Patients With Type 2 Diabetes
Brief Title: Effect of a Combined Exercise Program on Neuropathic Pain and Perceived Quality of Life in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Gabriela Aké Palomo (Other)
Collaborators: Universidad Autónoma de Yucatán (Other)
Responsible Party: Sponsor-Investigator, Maria Gabriela Aké Palomo, Maria Gabriela Aké Palomo, Universidad Autónoma de Yucatán
Organization: Universidad Autónoma de Yucatán (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Folio No. 06-2022
Record Dates: First submitted 2022-12-05; First posted 2023-01-27 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2; Neuropathic Pain; Neuropathy, Diabetic
Keywords: Diabetes Mellitus type 2; Neuropathic pain; combined exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Neuralgia; Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: A prospective, longitudinal, quasi-experimental study of repeated measures (pretest-posttest)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined Exercise (Experimental): Therapeutic exercise program
  Interventions: Other: Combined Exercise

INTERVENTIONS:
Other: Combined Exercise — Therapeutic exercise program will be applied that will include two modalities: aerobic and resistance exercise. The duration will be 8 weeks with a frequency of 3 sessions per week, with a duration per session of 60 minutes.

SUMMARY:
Therapeutic exercise is one of the therapies used as a treatment for diabetic neuropathy, which is a complication of diabetes. In order to reduce pain and improve the perception of quality of life, a combined therapeutic exercise program will be implemented as an adjuvant and non-pharmacological treatment for diabetic neuropathy.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, quasi-experimental study of repeated measures (pretest-posttest), has been approved by the research and ethics committee of the Faculty of Medicine of the Autonomous University of Yucatan, issuing a report on October 26, 2022. An identification form will be filled out that will include socio-demographic and clinical data: presence of type II diabetes, presence of neuropathy, sex, age, marital status, schooling, occupation, BMI, time of diagnosis, HbA1C, insulin use, medical treatment and a neurological examination of the extremities. The DN4 questionnaire will be used to evaluate neuropathic pain and its characteristics, the VAS will be used to evaluate the degree of intensity or severity of pain, and the SF-36 questionnaire will be used to evaluate perception before and after the combined exercise program. During the intervention stage, a therapeutic exercise program will be applied that will include two modalities: aerobic and resistance exercise in the facilities of the Unidad Universitaria de Inserción social de San José Tecoh. The duration will be 8 weeks with a frequency of 3 sessions per week, with a duration per session of 60 minutes each, to achieve the minimum total time suggested by the guidelines of 150 minutes per week. These exercises will be prescribed in three phases to increase times, series, repetitions and resistances in a progressive manner according to the Borg scale. For the analysis of the variables, the parametric Student's t-test for related samples or the nonparametric Wilcoxon test with significance at 95% reliability will be used. The implementation of the study can demonstrate significant improvements in the symptomatology of diabetic neuropathy, directly impacting on the perception of the quality of life of patients with type II diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes type 2
* Patients with neuropathy
* Patients with medical treatment

Exclusion Criteria:

* Patients with several limit function
* Patients with foot ulcer or amputation
* Patients who are involved in a exercise program already

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in neuropathic pain on Douleur Neuropathique-4 (DN4) at 8 weeks | Baseline and week 8
  The DN4 questionnaire will be used to evaluate neuropathic pain and its characteristics. DN4 for neuropathic pain consists of interview questions and physical tests. It has 10 items grouped into four questions: seven items relating to the pain description (burning, painful cold, electric shocks) and to its associated abnormal sensations (tingling, pins and needles, numbness, itching), and the other three items relating to a brief bedside neurological examination in the painful area (touch hypoaesthesia, pinprick hypoaesthesia and tactile dynamic allodynia). For scoring, 1 is given to each positive and 0 to each negative item (total score range 0-10). The cut-off value for diagnosis of neuropathic pain is a total score of 4.
Change from baseline in pain intensity on Visual Analogue Scale (VAS) at 8 weeks | Baseline and week 8
  Pain severity will be assessed using VAS. Each patient will be asked to choose in a perpendicular line on the VAS at the point that signifies the pain severity. The score is ranged 0-10, 0 suggests no pain and 10 suggest severe pain.
Change from baseline in quality of life on the short form-36 questionnaire (SF-36) at 8 weeks | Baseline and week 8
  The 36-item questionnaire consists of eight domains (general health, mental health, role emotion, role physical, body pain, social function, physical function and vitality), which can be further aggregated into a physical component score (PCS) and mental component score (MCS). Total score ranges from 0 to 100, 0 indicates the poor quality of life and 100 indicates the best quality of life.

SECONDARY OUTCOMES:
Socio-demographic data | Before intervention
  An identification form will be filled out at the beginning of the study that will include socio-demographic information: sex (woman/man), age (years), marital status (single/married/widowed/divorced), educational stage (Primary education/High School/University/Master) and occupation (yes/no). All data will be presented in frequency and percentage.
Clinical data | Before intervention
  An identification form will be filled out at the beginning of the study that will include clinical information: presence of type II diabetes, presence of neuropathy, time of diagnosis (years), Glycemic status (A1C percentage), insulin use (yes/no) and medical treatment. All data will be presented in frequency and percentage.
  For the neurological examination of the extremities, three instruments will be used: the 10g or Semmes-Weinstein monofilament, 128 hertz tuning fork and Taylor reflex hammer.
Weight measurement | Before intervention
  Body weight will be measured in kilograms (kg) using the body weight scale "Omron HBF-514C".
Height measurement | Before intervention
  Height will be measured in meters (m) using a stadiometer.
Body Mass Index (BMI) measurement | Before intervention
  BMI will be calculated by dividing the weight in kilograms by the height in metres squared (kg/m^2).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gabriela Aké Palomo, Principal Investigator — Facultad de Medicina; Damaris Francis Estrella Castillo, PhD, Study Director — Falcultad de Medicina; Gloria de los Ángeles Uicab Pool, PhD, Study Director — Facultad de Enfermeria; Hector Armado Rubio Zapata, Study Director — Facultad de Medicina
Locations (1):
- Unidad Universitaria de Inserción Social San José Tecoh, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pop-Busui R, Boulton AJ, Feldman EL, Bril V, Freeman R, Malik RA, Sosenko JM, Ziegler D. Diabetic Neuropathy: A Position Statement by the American Diabetes Association. Diabetes Care. 2017 Jan;40(1):136-154. doi: 10.2337/dc16-2042. No abstract available. PMID 27999003
- [Background] Scholz J, Finnerup NB, Attal N, Aziz Q, Baron R, Bennett MI, Benoliel R, Cohen M, Cruccu G, Davis KD, Evers S, First M, Giamberardino MA, Hansson P, Kaasa S, Korwisi B, Kosek E, Lavand'homme P, Nicholas M, Nurmikko T, Perrot S, Raja SN, Rice ASC, Rowbotham MC, Schug S, Simpson DM, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ, Barke A, Rief W, Treede RD; Classification Committee of the Neuropathic Pain Special Interest Group (NeuPSIG). The IASP classification of chronic pain for ICD-11: chronic neuropathic pain. Pain. 2019 Jan;160(1):53-59. doi: 10.1097/j.pain.0000000000001365. PMID 30586071
- [Background] Perez C, Galvez R, Huelbes S, Insausti J, Bouhassira D, Diaz S, Rejas J. Validity and reliability of the Spanish version of the DN4 (Douleur Neuropathique 4 questions) questionnaire for differential diagnosis of pain syndromes associated to a neuropathic or somatic component. Health Qual Life Outcomes. 2007 Dec 4;5:66. doi: 10.1186/1477-7525-5-66. PMID 18053212
- [Background] Pereira EV, Tonin FS, Carneiro J, Pontarolo R, Wiens A. Evaluation of the application of the Diabetes Quality of Life Questionnaire in patients with diabetes mellitus. Arch Endocrinol Metab. 2020 Feb;64(1):59-65. doi: 10.20945/2359-3997000000196. Epub 2020 Mar 13. PMID 32187271
- [Background] Kanaley JA, Colberg SR, Corcoran MH, Malin SK, Rodriguez NR, Crespo CJ, Kirwan JP, Zierath JR. Exercise/Physical Activity in Individuals with Type 2 Diabetes: A Consensus Statement from the American College of Sports Medicine. Med Sci Sports Exerc. 2022 Feb 1;54(2):353-368. doi: 10.1249/MSS.0000000000002800. PMID 35029593
- [Result] Pan B, Ge L, Xun YQ, Chen YJ, Gao CY, Han X, Zuo LQ, Shan HQ, Yang KH, Ding GW, Tian JH. Exercise training modalities in patients with type 2 diabetes mellitus: a systematic review and network meta-analysis. Int J Behav Nutr Phys Act. 2018 Jul 25;15(1):72. doi: 10.1186/s12966-018-0703-3. PMID 30045740